CLINICAL TRIAL: NCT05968794
Title: The Effectiveness of Cerclage for the Reduction of Extreme Preterm Birth and Perinatal Mortality in Twin Pregnancies With a Short Cervix or Dilatation
Brief Title: Cerclage for the Reduction of Extreme Preterm Birth in Twin Pregnancies With a Short Cervix or Dilatation
Acronym: TWIN Cerclage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Martijn A. Oudijk, MD, PhD, Prof.dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TwinC
Record Dates: First submitted 2023-04-22; First posted 2023-08-01 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Twin pregnancy; Cerclage
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: International, multicenter randomized controlled trial
Masking Description: Participants and investigators will not be blinded for the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerclage (Experimental): A vaginal cerclage is a short and minor surgical procedure performed under general or regional anesthesia. An unabsorbable suture is placed around/through the cervix to close the cervical canal and to increase its firmness, in order to reduce cervical insufficiency.
  Interventions: Procedure: Vaginal cerclage
- Standard care (No Intervention): The comparator will be standard treatment according to the current Dutch (NVOG) guideline from 2018, which is to not perform or offer an intervention such as vaginal cerclage. This is in line with the standard care in the participating hospitals in Belgium.

INTERVENTIONS:
Procedure: Vaginal cerclage — A vaginal cerclage is a short and minor surgical procedure performed under general or regional anesthesia. An unabsorbable suture is placed around/through the cervix to close the cervical canal and to increase its firmness, in order to reduce cervical insufficiency.
  Arms: Cerclage

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of a cerclage in women with a twin pregnancy with a midpregnancy short cervix or cervical dilatation compared to standard treatment (no cerclage) in the prevention of extreme preterm birth < 28 weeks of gestational age.

The main question it aims to answer is: What is the effectiveness of a cerclage in women with a twin pregnancy with a midpregnancy short cervix or cervical dilatation compared to standard treatment (no cerclage) in the prevention of extreme preterm birth < 28 weeks of gestational age?

Participants will be randomly assigned to the intervention (cerclage) or comparison (no cerclage) group.

DETAILED DESCRIPTION:
Rationale: In the Netherlands, 250 women with a twin pregnancy deliver at < 28 weeks per year, resulting in 157 perinatal deaths. A vaginal cerclage could be an effective surgical method to reduce cervical insufficiency and with that preterm birth, but the evidence regarding its effectiveness on extreme preterm birth and (long term) neonatal outcome is lacking.

Objective: To assess the effectiveness of a cerclage in women with a twin pregnancy with a midpregnancy short cervix or cervical dilatation compared to standard treatment (no cerclage) in the prevention of extreme preterm birth < 28 weeks of gestational age.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: A vaginal cerclage is a minor and safe surgical procedure commonly performed in singleton pregnancies with a short cervix and a previous preterm birth in all the participating centers, thus there is experience in the participating hospitals. The results of this study will show whether a vaginal cerclage reduces extreme preterm birth in women with twin pregnancy and a short cervix, and its accompanying perinatal complications. If proven effective, the implementation of this intervention will have a huge impact on the lifelong health of these children and their families.

ELIGIBILITY:
Inclusion Criteria: Women (> 16 years of age) with a twin pregnancy and:

* an asymptomatic short cervix at routine ultrasound investigation (below 24 weeks of gestation) OR
* cervical dilatation (below 24 weeks of gestation)

Exclusion Criteria:

* Women with a mono-amniotic twin pregnancy
* Women with twin pregnancy in which one or both children are diagnosed with a major structural, congenital or chromosomal abnormality that is likely to influence the composite adverse neonatal outcome.
* Women with dilatation of the cervix and signs of clinical intra-uterine infection, defined by the presence of fever ≥ 38 degrees Celsius.
* Women with overt symptoms of preterm labour at time of measurement of short cervix (regular contractions, PPROM, recurrent blood loss).
* Women with a placenta previa, defined as a placenta position covering the internal ostium of the cervix.
* Women who do not master the Dutch of English language and therefore not able to give written consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of extreme preterm birth | <28 weeks of gestation

SECONDARY OUTCOMES:
Rate of Preterm birth | <24, <32, <34 and <37 weeks
  Indicated and spontaneous
Rate of Premature rupture of membranes | Up to 42 weeks of pregnancy
Gestational age at delivery | At delivery
Days on ventilation support | Up to 3 months corrected age
  Neonatal
Days in NICU | Up to 3 months corrected age
  Neonatal
Maternal quality of life assessed by the 'European Quality of life 5-Dimension 5-Level' score | Up to 3 months corrected age
  The 'European Quality of life 5-Dimension 5-Level' score consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) that are rated using five levels (no problems (1), slight problems (2), moderate problems (3), severe problems (4), extreme problems (5)). A unique health state is defined by combining one level from each of the five dimensions. Each state is referred to by a 5-digit code, The best score is 11111 and the worst score is 55555.
Rate of maternal outcomes | Up to 3 months corrected age
  Sepsis, need for antibiotics, need to remove cerclage in operation room, mode of delivery (% caesarean delivery).
Adverse neonatal outcome | Up to 3 months corrected age
  A composite for adverse neonatal outcome (including bronchopulmonary dysplasia, periventricular leucomalacia > grade 1, intraventricular hemorrhage > grade 2, necrotizing enterocolitis > stage 2, retinopathy of prematurity > stage 2, proven sepsis and perinatal death)
Number of neonates with bronchopulmonary dysplasia | Up to 3 months corrected age
Number of neonates with periventricular leucomalacia > grade 1 | Up to 3 months corrected age
Number of neonates with intraventricular hemorrhage > grade 2 | Up to 3 months corrected age
Number of neonates with necrotizing enterocolitis > stage 2 | Up to 3 months corrected age
Number of neonates with retinopathy of prematurity > stage 2 | Up to 3 months corrected age
Number of neonates with proven sepsis | Up to 3 months corrected age
Perinatal death | Up to 3 months corrected age

OTHER OUTCOMES:
Healthcare costs assessed by the 'iMTA Medical Consumption Questionnaire' | Up to one week after labour and up to 3 months corrected age
  Costs will be measured from a societal perspective using a web-based questionnaires based on the 'iMTA Medical Consumption Questionnaire'. The scoring involves quantifying the reported healthcare resource use based on the responses provided by the participants. The questionnaire collects information about various types of healthcare services and resources, such as hospitalizations, outpatient visits and medication use.
Healthcare costs assessed by the 'iMTA Productivity Cost Questionnaire' | Up to one week after labour and up to 3 months corrected age
  Costs will be measured using a web-based questionnaires based on the 'iMTA Productivity Cost Questionnaire'. It collects information on the duration and frequency of productivity loss, as well as associated costs.The questionnaire consists of multiple sections and items that gather data on work-related activities, job characteristics, and productivity impact. Respondents are asked to report on their own productivity or that of a specific population (e.g., patients, caregivers) over a defined period.

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (5):
  - University Medical Center Antwerpen, Antwerp
  - University Medical Center Sint-Lucas Brugge, Bruges
  - Hospital Oost-Limburg Genk, Genk
  - University Medical Center Gent, Ghent
  - University Medical Center Leuven, Leuven
- Netherlands (8):
  - University Medical Center Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - University Medical Center Leiden, Leiden
  - University Medical Center Maastricht, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Centre, Rotterdam
  - University Medical Center Utrecht, Utrecht
  - Maxima Medical Centre, Veldhoven

IPD SHARING:
Plan to Share IPD: Yes
The manuscript will be published in an Open Access journal that provides a PID (e.g., a DOI or URN)
Supporting Information: Study Protocol

REFERENCES:
- [Derived] van Gils L, de Boer MA, Bosmans J, Duijnhoven R, Schoenmakers S, Derks JB, Prins JR, Al-Nasiry S, Lutke Holzik M, Lopriore E, van Drongelen J, Knol MH, van Laar JOEH, Jacquemyn Y, van Holsbeke C, Dehaene I, Lewi L, van der Merwe H, Gyselaers W, Obermann-Borst SA, Holthuis M, Mol BW, Pajkrt E, Oudijk MA. Study protocol for two randomised controlled trials evaluating the effects of Cerclage in the reduction of extreme preterm birth and perinatal mortality in twin pregnancies with a short cervix or dilatation: the TWIN Cerclage studies. BMJ Open. 2024 May 10;14(5):e081561. doi: 10.1136/bmjopen-2023-081561. PMID 38729756